CLINICAL TRIAL: NCT06358339
Title: The Tailored Evidence-based Enhancements in Mental Health-Gamified and Individualized Follow-Up Treatment for Suicide (TEEM-GIFTS) : Implementing a Gamified MHealth Intervention to Reduce Post-Discharge Suicide Risk in Patients with Mental Disorders Using Multiphase Optimization Strategy (MOST)
Brief Title: TEEM-GIFTS: a Gamified MHealth to Reduce Post-Discharge Suicide Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Kangning Hospital (Other)
Responsible Party: Principal Investigator, Fengsu Hou, Research Associate Professor, Shenzhen Kangning Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 72374095
Record Dates: First submitted 2024-03-20; First posted 2024-04-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Suicide
Keywords: Psychiatric patients; Post-discharge suicide; Gamification; Multiphase optimization strategy; Implementation science
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group. At the confirmation phase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group. At the confirmation phase, participants will be assigned into Group 17 to Group 18 randomly, with 160 participants in each group.
Who Masked: Participant, Investigator
Masking Description: After recruitment and the baseline survey, participants will be assigned into Group 1 to Group 16 by simple randomization in R program. The allocation ratio in randomization will be 1:1. Participants, LHSs, nurses who perform recruitment and baseline survey, and investigators who perform follow-ups will be blinded to the assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (18):
- Routine Tracker, Mind Care, Social Connectivity, and Achievement & Rewards (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group.
  The TEEM app with the intervention condition of Routine Tracker, Mind Care, Social Connectivity, and Achievement & Rewards.
  Interventions: Other: TEEM
- Routine Tracker, Mind Care and Social Connectivity (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group.
  The TEEM app with the intervention condition of Routine Tracker, Mind Care and Social Connectivity.
  Interventions: Other: TEEM
- Routine Tracker, Social Connectivity, and Achievement & Rewards (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group.
  The TEEM app with the intervention condition of Routine Tracker, Social Connectivity, and Achievement & Rewards.
  Interventions: Other: TEEM
- Routine Tracker and Achievement & Rewards (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group.
  The TEEM app with the intervention condition of Routine Tracker and Achievement & Rewards.
  Interventions: Other: TEEM
- Routine Tracker and Social Connectivity (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group.
  The TEEM app with the intervention condition of Routine Tracker and Social Connectivity.
  Interventions: Other: TEEM
- Routine Tracker and Mind Care (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group.
  The TEEM app with the intervention condition of Routine Tracker and Mind Care.
  Interventions: Other: TEEM
- Routine Tracker and Achievement & Reward (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group.
  The TEEM app with the intervention condition of Routine Tracker and Achievement & Reward.
  Interventions: Other: TEEM
- Routine Tracker (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group.
  The TEEM app with the intervention condition of Routine Tracker only.
  Interventions: Other: TEEM
- Mind Care, Social Connectivity, and Achievement & Rewards (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group.
  The TEEM app with the intervention condition of Mind Care, Social Connectivity, and Achievement & Rewards.
  Interventions: Other: TEEM
- Mind Care and Social Connectivity (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group
  The TEEM app with the intervention condition of Mind Care and Social Connectivity.
  Interventions: Other: TEEM
- Mind Care and Achievement & Rewards (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group.
  The TEEM app with the intervention condition of Mind Care and Achievement & Rewards.
  Interventions: Other: TEEM
- Mind Care (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group.
  The TEEM app with the intervention condition of Mind Care only.
  Interventions: Other: TEEM
- Social Connectivity and Achievement & Rewards (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group.
  The TEEM app with the intervention condition of Social Connectivity and Achievement & Rewards.
  Interventions: Other: TEEM
- Social Connectivity (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group.
  The TEEM app with the intervention condition of Social Connectivity only.
  Interventions: Other: TEEM
- Achievement & Rewards (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group.
  The TEEM app with the intervention condition of Achievement & Rewards only.
  Interventions: Other: TEEM
- Brief contact intervention (Experimental): At the optimization phrase, participants will be assigned into Group 1 to Group 16 randomly, with 20 participants in each group.
  Participants will receive care as usual (receiving brief contact intervention which mention in the study NCT04907669)
  Interventions: Other: TEEM
- Optimized TEEM (Experimental): At the confirmation phase, participants will be assigned into Group 17 to Group 18 randomly, with 160 participants in each group.
  The TEEM app with the optimized intervention condition from the optimization phase.
  Interventions: Other: TEEM
- Care as usual (Experimental): At the confirmation phase, participants will be assigned into Group 17 to Group 18 randomly, with 160 participants in each group.
  Participants will receive care as usual (receiving brief contact intervention which mention in the study NCT04907669)
  Interventions: Other: TEEM

INTERVENTIONS:
Other: TEEM — The TEEM app will provide four types of gamified intervention elements as Routine Tracker, Mind Care, Social Connectivity, and Achievement & Rewards which providing services including brief contact intervention, mCBT, health education, venting space, mood sharing, etc. Only enrolled participants have access to log in and use the app.

SUMMARY:
Patients with mental disorders are at significantly higher risk of suicide after discharge compared to the general population and patients with other diseases. Currently, there is a lack of post-discharge community suicide risk management services in China. The research team's preliminary research suggests that mHealth interventions are well-accepted and feasible for reducing the suicide risk in patients with mental disorders. Furthermore, the inclusion of gamification elements can enhance treatment adherence and user engagement. However, determining the appropriate combination of gamification elements and evaluating the implementation effectiveness of gamified mHealth interventions for suicide risk are challenges in transforming these into regular community mental health services. This study will leverage gamification theory and community-based participatory research to design a gamified mHealth intervention model aimed at reducing suicide risk among discharged patients with mental disorders, and to develop a corresponding management strategy. Using the multi-phase optimization strategy (MOST), the study will identify the optimal combination of gamification elements to reduce suicide risk and increase the outpatient follow-up rate. Through an implementation science framework, the investigators will evaluate the process, outcomes, cost, and feasibility of this management strategy with the goal of reducing suicide risk among these patients. The findings from this study will provide a scientific basis for innovative suicide risk management models for discharged patients with mental disorders in China, thereby paving the way for the application of implementation science in mental health.

DETAILED DESCRIPTION:
The Tailored Evidence-based Enhancements in Mental health (TEEM) projects, adhering to implementation science principles, encompass various studies aimed at improving mental health care in China. Among these is the Gamified and Individualized Follow-Up Treatment for Suicide (GIFTS) study. Based on the multi-phase optimization strategy (MOST), this is a mixed-methods study with three phases. The selection phase involves forming the gamified mHealth suicide risk management strategy and system through community participatory research. The optimization phase involves testing and adjusting the intervention elements for the gamified mHealth strategy through a factorial design randomized controlled trial (RCT) to evaluate the effectiveness of different combinations of intervention elements in reducing suicide risk. The confirmation phase will assess the optimized strategy based on the Implementation Outcomes Framework (IOF), focusing primarily on patient outcomes obtained through a standard RCT.

1. Selection phase Based on literature review, the research team has identified several gamification elements, including avatar, points, badges, missions, level & leaderboards, team mates & team missions, venting space, mood sharing, achievement and titles, and rewards, etc. During developing the gamification mHealth app (TEEM), the investigators categorize the elements into four types of intervention elements as Routine Tracker, Mind Care, Social Connectivity, and Achievement & Rewards; meanwhile, under the community-based participatory research (CBPR) framework, the investigators aim to explore the appropriate content of gamification mHealth interventions, the acceptance and feasibility of such interventions among discharged psychiatric patients, as well as structural and perceptual barriers during implementation.

   In specific, the research team will recruit discharged patients with mental disorders and their lay health care supporters (LHSs) who are usually their family members, psychiatrists and nurses, psycho-crisis intervention team members, community mental health workers and mental health social workers as the community team, and will categorize the community team into three sub-groups, the patients-LHSs group, the clinic mental health service provider group (psychiatrists and nurses, and psycho-crisis intervention team members), and the community mental health service provider group (community mental health workers and mental health social workers). The investigators will conduct three focus group interviews in each sub-group and ten to fifteen cases of individual in-depth interview with the community to avoid bias in focus groups and to protect privacy related to personal experience in suicide and suicide intervention. There will be scheduled meetings with the community to discuss and revise the intervention strategy before implementation. Purposive sampling will be applied to recruit participants for the community team. For each type of sub-group, there will be five to eight members
2. Optimization phase The research team will conduct a a factorial design randomized controlled trial (RCT) to evaluate the effectiveness of different combinations of intervention elements in reducing suicide risk. There are four intervention elements as mentioned, thus there will be 16 groups in the factorial design RCT. The research team will recruit discharged patients with mental disorders from Shenzhen Mental Health Center/Shenzhen Kangning Hospital (SKH).

   The research team sets the standard for optimizing interven elements as follows: The experimental group implementing the intervention element and the experimental group not implementing the intervention element should have an effect difference in reducing the suicide risk by 35%, which will be used as the basis for calculating the sample size of this study. This study aims to detect a 35% difference (δ) in the implementation of the intervention elements with a test level of α=0.05 and a test power (1-β) of 80%. A total of 260 patients need to be recruited for this study. Assuming a loss to follow-up rate of 20% and considering the number of experimental groups, the final sample size is 320 patients.

   In accordance with the factorial design, the optimization phase will consist of 16 groups, and this is due to the four types of intervention elements and their 16 possible intervention conditions. Thus, after recruitment and the baseline survey, participants will be assigned into Group 1 to Group 16 by simple randomization in R program, with 20 participants in each group. Further, participants in each group will only have access to a single intervention condition of elements assigned to their group. Noted, the intervention app TEEM will be developed during the selection phase, and there will be an Android/iOS version of TEEM and a mini-program in the WeChat platform. Participants, LHSs, nurses who perform recruitment and baseline survey, and investigators who perform follow-ups will be blinded to the assignment.

   To evaluate post-discharge suicide risk more cautiously and to provide crisis intervention in time, face-to-face interview will be conducted to collect information. Trained nurses in SKH will recruit participants and perform baseline survey. The research assistants will contact participants, schedule visits to SKH out-patient clinics , and complete follow-up questionnaires after out-patient visits at one week, one month, and three months after discharge. If participants refused subsequent visits, the investigators would schedule home visits to complete the survey by research assistants and community mental health workers. The condition that resulted in the greatest decrease in participants' suicide risk three months after discharge is the optimized intervention condition.
3. Confirmation phase This phase will assess the optimized intervention, focusing primarily on patient outcomes obtained through a standard RCT, in which intervention group (Group 17) will receive the optimized intervention condition and the control group (Group 18) will receive care as usual. Similar to the optimization phase, the research team will recruit discharged patients with mental disorders from SKH. The sample size (n=320) and randomization process will be consistent with optimization phase. Data collection, baseline survey and follow-up schedule are similar to the optimization phase. The primary outcomes are suicide risk and the rate of re-visits to outpatient clinic at three months after discharge. Secondary outcomes will be illustrated later in the Outcome measures section.
4. Study outcomes and measurements The implementation outcomes of the overall project are based on the Implementation Outcomes Framework, in which detailed primary and secondary outcomes of the study will be collected at 3 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

For patients

* Being 18 years and above;
* Being diagnosed with mental disorders;
* Having received inpatient care for three days or more;
* Living in Shenzhen and having no plan to leave Shenzhen in the following 12 months after discharge;
* Being able to use apps or WeChat (WeChat mini program) on smart phones.

For lay health care supporters (LHSs)

* Being 18 years and above;
* Being without any diagnosis of mental disorder;
* Being the lay health care supporter in the family;
* Living in Shenzhen and having no plan to leave Shenzhen in the following 12 months after discharge;
* Being able to use apps or WeChat (WeChat mini program) on smart phones.

For the clinic and community mental health service providers

* Being 18 years and above;
* Having practiced in mental health service at least for 12 months.

Exclusion criteria For patients

* Refusing to provide written consent or be unable to provide written consent due to any cognitive problems.
* Being discharged by the patient's or LHSs' demand against medical advice.
* With no ID, no stable residence nor any source of income.

For For lay health care supporters (LHSs)

* Refusing to provide written consent.

For the clinic and community mental health service providers

* Refusing to provide written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Suicide ideation at three months after discharge | It will be evaluated at one week, one months and three months after discharge.
  This study will use the Beck Suicide Ideation Scale-Chinese Version (BSI-CV) to assess participants' suicide ideation. The BSI-CV includes 19 items, and each item scores from 0 to 2 with a total score ranging from 0 to 38, and a higher score indicates a higher level of suicide ideation. The total score and its trajectory from baseline to three months after discharge will be recorded and compared.
The rate of re-visits to outpatient clinic at three months after discharge | It will be evaluated at one week, one months and three months after discharge.
  Responses to the question "How many times have you re-visited the outpatient clinic at SKH in the past three months? " will be recorded and compared. In clinic, patients must visit the outpatient clinic one week post-discharge to refill their medication, which can only be prescribed for a maximum of 30 days, resulting in at least four subsequent visits to the clinic. Thus, we define the rate of outpatient clinic revisits as the number of participants who complete all revisits divided by the total number of participants.

SECONDARY OUTCOMES:
Self-determination at at three months after discharge | It will be evaluated at one week, one months and three months after discharge.
  This study will use the Self-Determination Scale-Chinese Version (SDS) to assess participants' the level of self-determination. The SDS includes 10 items, and each item includes two statements, with scoring options ranging from 'agree only with statement A' to 'agree only with statement B' on a scale of 1-9 with a total score ranging from 10 to 90, and a higher score indicates a higher level of self-determination. The total score and its trajectory from baseline to three months after discharge will be recorded and compared.
Social connectedness at three month after discharge | It will be evaluated at one week, one months and three months after discharge.
  Social connectedness will be measured by the Social Connectedness Scale (SCS) to evaluate participants' social connected ness after discharge. The SCS is a 20-item scale, and each item is on a 6-Likert continuum (from "Strongly disagree" to "Strongly agree") scoring from 1 to 6. A higher total score indicates a higher level of social connectedness. The total score and its trajectory from baseline to three months after discharge will be recorded and compared.
Social support at three months after discharge | It will be evaluated at one week, one months and three months after discharge.
  Social support will be measured by the 23-item Duke Social Support Index (DSSI) to evaluate participants' social support after discharge. The DSSI investigates social support by social interaction, perceived social support and instrumental social support. Every answer has been assigned a score, and the total reflects the sum of the items ranging from 11 to 45. A higher total score indicates a higher level of social support. The total score and its trajectory from baseline to three months after discharge will be recorded and compared.

OTHER OUTCOMES:
Times of re-hospitalization for mental disorders | It will be evaluated at one week, one months and three months after discharge.
  Responses to the question "How many times have you been hospitalized for mental disorders" will be recorded and compared.
Attitudes towards the acceptability of the intervention | It will be evaluated by three focus group interviews immediately after the confirmation phase, and each interview will be about 60 to 120 minutes.
  This is a mixed methods study, and the investigators will conduct community-based participatory research (CBPR) to evaluate the implementation of the intervention. After the confirmation phase, focus group interviews will be conducted with the CBPR team understand the community's attitudes towards the acceptability of the intervention. Of note, participants (the patients, LHSs, clinical and community mental health providers) are recruited for the qualitative interviews only, who are different from the MOST phases.
Attitudes towards the adoption of the intervention | It will be evaluated by three focus group interviews immediately after the confirmation phase, and each interview will be about 60 to 120 minutes.
  This is a mixed methods study, and the investigators will conduct community-based participatory research (CBPR) to evaluate the implementation of the intervention. After the confirmation phase, focus group interviews will be conducted with the CBPR team understand the community's attitudes towards the adoption of the intervention. Of note, participants (the patients, LHSs, clinical and community mental health providers) are recruited for the qualitative interviews only, who are different from the MOST phases.
The adoption rate of the intervention in patients | It will be evaluated at three months after discharge.
  The rate will be measured by the number of participants who use the TEEM app divided by the number of participants at the end of the study. Of note, this outcome evaluates the implementation process of the intervention.
Attitudes towards the equity of the intervention | It will be evaluated by three focus group interviews immediately after the confirmation phase, and each interview will be about 60 to 120 minutes.
  This is a mixed methods study, and the investigators will conduct community-based participatory research (CBPR) to evaluate the implementation of the intervention. After the confirmation phase, focus group interviews will be conducted with the CBPR team understand the community's attitudes towards the equity of the intervention. Of note, participants (the patients, LHSs, clinical and community mental health providers) are recruited for the qualitative interviews only, who are different from the MOST phases.
Attitudes towards the feasibility of the intervention | It will be evaluated by three focus group interviews immediately after the confirmation phase, and each interview will be about 60 to 120 minutes.
  This is a mixed methods study, and the investigators will conduct community-based participatory research (CBPR) to evaluate the implementation of the intervention. After the confirmation phase, focus group interviews will be conducted with the CBPR team understand the community's attitudes towards the feasibility of the intervention. Of note, participants (the patients, LHSs, clinical and community mental health providers) are recruited for the qualitative interviews only, who are different from the MOST phases.
Attitudes towards the patient-centeredness of the intervention | It will be evaluated by three focus group interviews immediately after the confirmation phase, and each interview will be about 60 to 120 minutes.
  This is a mixed methods study, and the investigators will conduct community-based participatory research (CBPR) to evaluate the implementation of the intervention. After the confirmation phase, focus group interviews will be conducted with the CBPR team understand the community's attitudes towards the patient-centeredness of the intervention. Of note, participants (the patients, LHSs, clinical and community mental health providers) are recruited for the qualitative interviews only, who are different from the MOST phases.
Cost for implementing the TEEM-GIFTS | It will be evaluated immediately after the confirmation phase.
  It will be measured by the overall cost on developing and implementing the TEEM during the study. Of note, this outcome evaluates the implementation process of the intervention.
Fidelity of the study | It will be evaluated immediately after the confirmation phase.
  The investigators will develop a checklist to evaluate the fidelity of the overall study. Of note, this outcome evaluates the implementation process of the intervention.
Efficiency of the intervention | It will be evaluated immediately after the confirmation phase.
  During the confirmation phase, the investigators will record the response speed of the app as experienced by users of TEEM. This term refers to how quickly an application reacts to user inputs or requests. It's a critical aspect of user experience, encompassing everything from tapping a button, swiping through content, to executing a command. Of note, this outcome evaluates the implementation process of the intervention.
Attitudes towards the safety of the intervention | It will be evaluated by three focus group interviews immediately after the confirmation phase, and each interview will be about 60 to 120 minutes.
  This is a mixed methods study, and the investigators will conduct community-based participatory research (CBPR) to evaluate the implementation of the intervention. After the confirmation phase, focus group interviews will be conducted with the CBPR team understand the community's attitudes towards the safety of the intervention. Of note, participants (the patients, LHSs, clinical and community mental health providers) are recruited for the qualitative interviews only, who are different from the MOST phases.
The timeliness of the intervention | It will be evaluated immediately after the confirmation phase.
  The investigators will record the time for the research team cost to response to participants' requests for crisis intervention and feedbacks.
Patients' perceived stigma from baseline to three months after discharge | It will be evaluated at one week, one months and three months after discharge.
  Perceived stigma will be evaluated the Chinese version of Link Perceived Devaluation-Discrimination Scale. The scale contains 12 items assessing the extent to which a person believes that other people will devalue or discriminate against someone with a mental illness. Each item is on a 4-Likert continuum (from "Strongly disagree" to "Strongly agree") scoring from 1 to 4. A higher total score indicates a higher level of perceived stigma. The total score and its trajectory from baseline to three months after discharge will be recorded and compared.
Patients' self-efficacy from baseline to three months after discharge | It will be evaluated at one week, one months and three months after discharge.
  Self-efficacy will be evaluated by the Chinese version of the General Self-Efficacy Scale. The scale contains 10 items, and each item is on a 4-Likert continuum (from "Not at all true" to "Exactly true") scoring from 1 to 4. A higher total score indicates a higher level of self-efficacy. The total score and its trajectory from baseline to three months after discharge will be recorded and compared.
Patients' compliance to treatment from baseline to three months after discharge | It will be evaluated at one week, one months and three months after discharge.
  Compliance to treatment will be evaluated by a 4-item self-administered questionnaire. The questionnaire inquires whether the patients take medications under the instruction on prescriptions (frequency, dosage, time, and selfdiscontinued medication). Each item is on a 4-Likert continuum (from "Not following the instruction" to "Exactly following the instruction") scoring from 1 to 4. A higher total score indicates a higher level of compliance to treatment. The total score and its trajectory from baseline to three months after discharge will be recorded and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Fengsu Hou, Ph.D., Principal Investigator — Shenzhen Kangning Hospital
Locations (1):
- Shenzhen Kangning Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Quantitative data will be publicly available through FigShare 12 months after the main studies are published in peer-reviewed journals. The data will contain deidentified demographic information, primary and secondary outcomes, and other covariate outcomes.
Supporting Information: Study Protocol
Time Frame: Twelve months after the main studies are published in peer-reviewed journals. The study protocol will be shared once published in peer-reviewed journal.
Access Criteria: Please contact the PI Fengsu Hou to request for the use of the data, and the requests should include detail contact information of applicants, the purpose of study, and the analysis plan.

REFERENCES:
- [Background] Sebastian Deterding, Dan Dixon, Rilla Khaled, and Lennart Nacke. 2011. From game design elements to gamefulness: defining
- [Background] Deci EL, Ryan RM, Handbook of self-determination research[M/OL]. Rochester, NY: University Rochester Press, 2002. https://psycnet.apa.org/record/2002-01702-000.
- [Background] Hopia H, Raitio K. Gamification in Healthcare: Perspectives of Mental Health Service Users and Health Professionals. Issues Ment Health Nurs. 2016 Dec;37(12):894-902. doi: 10.1080/01612840.2016.1233595. Epub 2016 Dec 1. PMID 27905826
- [Background] Christensen H, Farrer L, Batterham PJ, Mackinnon A, Griffiths KM, Donker T. The effect of a web-based depression intervention on suicide ideation: secondary outcome from a randomised controlled trial in a helpline. BMJ Open. 2013 Jun 28;3(6):e002886. doi: 10.1136/bmjopen-2013-002886. PMID 23811172
- [Background] Morris ZS, Wooding S, Grant J. The answer is 17 years, what is the question: understanding time lags in translational research. J R Soc Med. 2011 Dec;104(12):510-20. doi: 10.1258/jrsm.2011.110180. PMID 22179294
- [Background] Collins LM, Murphy SA, Nair VN, Strecher VJ. A strategy for optimizing and evaluating behavioral interventions. Ann Behav Med. 2005 Aug;30(1):65-73. doi: 10.1207/s15324796abm3001_8. PMID 16097907
- [Background] Collins LM, Baker TB, Mermelstein RJ, Piper ME, Jorenby DE, Smith SS, Christiansen BA, Schlam TR, Cook JW, Fiore MC. The multiphase optimization strategy for engineering effective tobacco use interventions. Ann Behav Med. 2011 Apr;41(2):208-26. doi: 10.1007/s12160-010-9253-x. PMID 21132416
- [Derived] Hou F, Liu H, Bai Y, Peng B, Chen G, Zhang Y, Wu D, Fu T, Hu L, Li J. Protocol of the Tailored Evidence-based Enhancements in Mental Health-Gamified and Individualized Follow-Up Treatment for Suicide (TEEM-GIFTS): a Multiphase Optimization Strategy (MOST) study implementing a gamified mHealth intervention to reduce postdischarge suicide risk in patients with mental disorders in Shenzhen. BMJ Open. 2025 Apr 15;15(4):e092339. doi: 10.1136/bmjopen-2024-092339. PMID 40233959